CLINICAL TRIAL: NCT07039409
Title: Effectiveness of Self-administered Acupressure Intervention in Managing Constipation of Adult Psychiatric Out-patient - A Pilot Study
Brief Title: Effectiveness of Self-administered Acupressure Intervention in Managing Constipation of Adult Psychiatric Out-patient
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Responsible Party: Principal Investigator, Dr Kelvin WONG Wai Kit, Assistant Professor, School of Nursing and Health Sciences, Hong Kong Metropolitan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIRB-2025-005-1
Record Dates: First submitted 2025-06-02; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Constipation; Psychiatric Drug Induced Constipation; Constipation Drug Induced
Keywords: constipation; psychiatric out-patient
MeSH Terms: conditions — Constipation | interventions — Acupressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): We will use the content-validated acupressure intervention used in our previous study [27]. The acupressure intervention will include the following five acupoints: Zhongwan (RN12), located on the upper abdomen and on the anterior midline 4 cun (just over 10 cm) above the centre of the umbilicus [15]; the right and left Tianshu (ST25), located in the central abdominal region and 2 cun (just over 5 cm) lateral to the umbilicus; and the right and left Quchi (LI11), located at the lateral end of the elbow crease when the forearm is bent and at the midpoint of the line connecting Chize (LU5) to the lateral epicondyle of the humerus.
  Interventions: Behavioral: Acupressure

INTERVENTIONS:
Behavioral: Acupressure — Patients will receive three 1-hour sessions of training at home within 3 days by Community Psychiatric Nurse (CPN), who was trained by an experienced TCM practitioner. They will learn acupressure. After the training, they will be assessed by the CPN to ensure that they are able to identify the acupoint based on reports of a sensation of obtaining 'Qi' when using the Point Locator device. They will then apply constant pressure for approximately 1 minute on each acupoint using the Acupen, as indicated by a marking in red by themselves. To ensure treatment compliance, the participants will apply this intervention once per day for 10 days. During the 10-day intervention period, and the patient should sign in on WhatsApp every day. If the patient is unable to use WhatsApp, the print edition of diary will be provided and supervision will be performed by short message and home visit during the 1st day, 5th day and 10th day of the intervention period.

SUMMARY:
Constipation is a common gastrointestinal condition characterised by unsatisfactory defecation as a result of infrequent stools, difficult stool passage or both. Overall, the average prevalence of constipation globally is estimated to be 16%. It affects approximately 14.3% of the population in Hong Kong. The condition incurs significant costs, with more than £162 million in associated costs in the UK National Health Service from 2017 to 2018. Similar expenses have been reported in Hong Kong and many Western countries. Previous studies have shown that constipation can lead to serious health complications, including paralytic ileus, faecal impaction, bowel obstruction and even premature death. It not only causes patient discomfort and reduces quality of life but also increases treatment costs.

Psychiatric patients, particularly those on psychotropic drugs such as antipsychotics and antidepressants, are more susceptible to constipation, with more than one third of such patients affected in Europe. This high prevalence may be due to the side effects of these drugs, as well as factors such as a sedentary lifestyle, negative symptoms of schizophrenia, a poor mental state, an unhealthy diet and insufficient fiber intake. The physical health of individuals with severe mental illness, including constipation, has become a major concern in recent years. However, the issues are often overlooked and under-researched, making their management a critical aspect of mental health care.

Common treatments for constipation include pharmacological and non-pharmacological interventions. While pharmacological interventions can effectively alleviate symptoms, they are short-term solutions. The long-term use of laxatives can cause serious side effects, such as bloating, allergic reactions, abdominal pain, metabolic disturbances and hepatotoxicity, which far outweigh the therapeutic effects. Alternative non-invasive interventions, such as auriculotherapy and behavioural therapy, have been found to be ineffective. Only one randomised controlled trial (RCT) of abdominal massage therapy in 60 older adults with constipation in Sweden showed decreased constipation severity and increased bowel movement frequency. However, this did not lead to a decrease in laxative intake, and the intervention requires a therapist to perform. These factors may reduce the accessibility and sustainability of the intervention. Therefore, the investigators propose to test a simpler and less expensive intervention to manage constipation in adult psychiatric out-patients. This intervention will incorporate the concept of self-help, acupressure.

Self-help concept: Since the 19th century, self-care has been a crucial element of healthcare systems. It is defined as a deliberate action undertaken by an individual to enhance their health or manage a disease. Florence Nightingale underscored the significance of personal hygiene and environmental factors in health, thereby establishing self-care as a fundamental principle in public health nursing. Orem further developed the notion of self-care, classifying it into three categories: universal self-care requisites, developmental self-care requisites and health-deviation self-care requisites. Barofsky divided self-care activities into four types: regulatory, preventive, reactive and restorative self-care. Both the World Health Organization and Pender accentuated the function of self-care in health enhancement, disease prevention and health restoration. In Orem's self-care model, patients perceived as active contributors to their own care.

Acupressure: Acupressure involves the application of constant pressure using a fingertip, thumb or the palm of the hand to specific acupoints to stimulate the flow of the life force known as 'Qi' in the meridians. In TCM, health problems are deemed to be due to pathogenic changes in Qi and an imbalance of 'Yin' and 'Yang'. Dysfunction of the viscera and bowels is induced by a deficiency or an excess of Qi in the body. Acupressure is based on the meridian theory, namely that Qi flows through the body along certain channels (meridians), which, if blocked, can cause illness. Stimulation at precise locations (acupoints) along these channels by a healthcare provider or the patients themselves can unblock the flow of Qi, relieving pain and restoring health. Acupressure is able to influence autonomic functions, which can affect the functioning of defecation. In addition, some studies have found that acupressure improves the symptoms of constipation in older adults and patients with stroke or with a vegetative status. Acupressure may have the positive effect of improving constipation. However, there have been no trials (RCTs or non-RCTs) assessing this in psychiatric out-patients. Therefore, the investigators propose to test the intervention in psychiatric out-patients.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong Chinese residents
2. Aged 18 or above
3. Meet the Rome III diagnostic criteria for constipation
4. Mentally stable and competent to perform self-care and learn acupressure, as recommended by their attending psychiatrists through letter/email
5. Able to understand the questionnaire and follow instructions for training

Exclusion Criteria:

1. Have an anatomical or physiological disorder of the gastrointestinal tract, such as malrotation, fistula or colonic neuropathy
2. Have a metabolic or endocrine disease
3. Have lead poisoning or vitamin D intoxication
4. Have had previous training in acupressure
5. Have a physical disability involving the upper limbs
6. Have planned surgery during the study period
7. Pregnant
8. receiving other kinds of "Qi" restoration-based treatment
9. Going to change medication or changed recently
10. Not in any other study or interventions that may improve constipation e.g. consulting dietitian, exercise programme etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Severity of constipation | Pre-intervention (Day1), Post-intervention(Day15)
  The Chinese version of the CAS (C-CAS) will be used to assess the severity of constipation symptoms. The 8-item C-CAS is commonly used and has a 3-point Likert scale, with ratings of '0 = no problem', '1 = some problems', and '2 = severe problems'. Higher total scores (possible range 0-16) indicate more severe symptoms.
Number of Complete Spontaneous Bowel Movements | Pre-intervention (Day1), Post-intervention(Day15)
  The number of complete spontaneous bowel movements (CSBMs) will be used to measure the severity of constipation symptoms which is recorded in the Bowel Movement Chart . According to a modification of the Rome II criteria, chronic functional constipation is defined as fewer than three CSBMs per week for more than 3 months. Therefore, more CSBMs per week indicates less-severe constipation symptoms.
Stool form | Pre-intervention (Day1), Post-intervention(Day15)
  Bristol Stool Form Scale (BSFS) will be used to measure symptom severity of constipation. The Bristol Stool Form Scale (BSFS), a graded visual scale of stool type from type 1 (hard lumps) to type 7 (watery diarrhea) which is recorded in the Patient's Bowel Movement chart, will be used to assess the patient's stool form.
Use of medication to relieve constipation symptoms | Pre-intervention (Day1), Post-intervention(Day15)
  A reduction in the use of medication (bulking agents, osmotic laxatives, stimulant laxatives, prokinetics and secretagogues) to relieve constipation symptoms

SECONDARY OUTCOMES:
Patients' quality of life | Pre-intervention (Day1), Post-intervention(Day15)
  The Chinese version of the PAC-QoL (C-PAC-QoL) will be used to assess specific disease-related patient quality of life. The PAC-QoL consists of 28 items categorised into four subscales, namely, dissatisfaction (five items), physical discomfort (four items), psychosocial discomfort (eight items) and worries and concerns (11 items). The items are rated on a 5-point Likert scale, ranging from '0 = none of the time or not at all' to '4 = all of the time or extremely'. A lower average total score indicates a higher health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Castle Peak Hospital, Tuenmen, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No